CLINICAL TRIAL: NCT06738433
Title: Efficacy and Tolerability of ABB I5 Prebiotic and ABB C22 Postbiotics for the Management of Constipation and Gastrointestinal Well-being: a Pilot Trial
Acronym: ABB i5/ABB C24
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: AB Biotek (Industry)
Collaborators: Grupo Colisée (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ABB i5/ABB C24
Record Dates: First submitted 2024-12-13; First posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Constipation
Keywords: constipation; prebiotic; postbiotic; gastrointestinal; dietary supplement
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ABB i5 (Experimental): Prebiotic ABB i5 (NextDext®, 5g)
  Interventions: Dietary Supplement: ABB i5
- ABB C24 (Experimental): ABB C24: Prebiotic ABB i5 (NextDext®, 5g) + yeast postbiotic ABB C22 (200 mg) in sachets containing 5,2 g
  Interventions: Dietary Supplement: ABB C24

INTERVENTIONS:
Dietary Supplement: ABB i5 — Prebiotic ABB i5 (NextDext®, 5g)
  Arms: ABB i5
Dietary Supplement: ABB C24 — ABB C24: Prebiotic ABB i5 (NextDext®, 5g) + yeast postbiotic ABB C22 (200 mg) in sachets containing 5,2 g
  Arms: ABB C24

SUMMARY:
In this study, we aim at assessing the benefits of dietary supplementation with ABB i5 and ABB C24, a combination of the the prebiotic ABB i5 and the postbiotic ABB C22, on the gut microbiota of people with constipation and on their gastrointestinal well-being.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who require hospitalization
* Constipation defined as the Rome IV criteria for constipation
* Patients with the ability to take the study product orally

Exclusion Criteria:

* History of allergy, idiosyncrasy, hypersensitivity or adverse reactions to the active principle or to any of the excipients.
* History or evidence of any medical conditions or medication used that, in the opinion of the principal investigator, could affect the safety of the subjects or interfere with the study evaluations
* Patients last palliative care en stage of "end of life" or "terminal"
* Amytriptilin (anti-depressive) and masalazine (anti-inflammatory) treatment
* Laxatives
* Antibiotic treatment in the previous 2 weeks
* Patients with IBS or any other gastrointestinal conditions that maybe the cause of the constipation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-04-25 (Actual); Primary Completion 2024-04-04 (Actual); Study Completion 2024-04-04 (Actual)

PRIMARY OUTCOMES:
Microbiota composition | from baseline to day 14 of supplementation
  Changes in microbiota composition through Shanon diversity test and statistical analyses (Continuous variables will be described as mean and standard deviation (SD) or as median and interquartile range; and categorical variables such as absolute frequencies and percentages).

SECONDARY OUTCOMES:
Transit time | from baseline to day 14 of supplementation
  transit time measured as methane on breathe testing
Tolerance and gastro-intestinal comfort | from baseline to day 14 of supplementation
  Tolerance and gastro-intestinal comfort (validated questionnaires) life questionnaire: the Digestion-associated Quality of Life Questionnaire (DQLQ)
Brain Derived Neurotrophic Factor (BDNF) | from baseline to day 14 of supplementation
  levels of Brain Derived Neurotrophic Factor (BDNF) (pg/mL)

CONTACTS AND LOCATIONS:
Locations (1):
- Isabel Roig, Barcelona, Barcelona, South Sudan

IPD SHARING:
Plan to Share IPD: Yes
Statistical results on microbiological data.
Supporting Information: Study Protocol
Time Frame: According to legislation

REFERENCES:
- [Derived] Culqui Levano DR, Rodriguez Sanz P, Palacios Sanchez R, Saldana Miranda MY, Santa Cruz Lopez CY, Mateus Rodriguez JA. Impact of prebiotics and postbiotics in the management of constipation: Analysis of their differentiated modulation of intestinal microbiota. Clin Nutr ESPEN. 2025 Oct;69:625-633. doi: 10.1016/j.clnesp.2025.08.003. Epub 2025 Aug 6. PMID 40780410